CLINICAL TRIAL: NCT00330837
Title: Ultrasound Scanning of Vascular Access Sites
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Other Study IDs: 0512116
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Catheterization, Central Venous; Ultrasonography

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Inadvertent puncture of an unintended object in a vascular access procedure is common and can lead to serious consequences. Inadvertent common carotid artery (CCA) puncture while targeting the internal jugular vein (IJV), for example, is reported to have an incidence of 2% - 8% and usually results in localized hematoma formation. The hematoma may enlarge rapidly if the patient is coagulopathic, or if a large puncture wound is produced by the introduction of the sheath itself into the CCA. Airway obstruction, pseudoaneurysm, arterio-venous fistula formation and retrograde aortic dissection have all been reported as a consequence of CCA puncture. In the presence of occlusive (atheromatous) carotid disease, inadvertent puncture may carry the risk of precipitating a cerebrovascular accident.

In this study, we aim to collect color Doppler and B-mode ultrasound videos from the most common ultrasound-guided vascular access sites - internal jugular vein, subclavian vein, femoral vein, basilic vein, and brachial vein. The videos will also include structures in close proximity to the intended veins. Using such database, we will run various vessel tracking and identification algorithms to evaluate their performance. Our ultimate goal is to develop an algorithm that will aid the ultrasound operator in identifying structures and differentiating between arteries and veins.

DETAILED DESCRIPTION:
Inadvertent puncture of an unintended object in a vascular access procedure is common and can lead to serious consequences. Inadvertent common carotid artery (CCA) puncture while targeting the internal jugular vein (IJV), for example, is reported to have an incidence of 2% - 8% and usually results in localized hematoma formation. The hematoma may enlarge rapidly if the patient is coagulopathic, or if a large puncture wound is produced by the introduction of the sheath itself into the CCA. Airway obstruction, pseudoaneurysm, arterio-venous fistula formation and retrograde aortic dissection have all been reported as a consequence of CCA puncture. In the presence of occlusive (atheromatous) carotid disease, inadvertent puncture may carry the risk of precipitating a cerebrovascular accident.

In this study, we aim to collect color Doppler and B-mode ultrasound videos from the most common ultrasound-guided vascular access sites - internal jugular vein, subclavian vein, femoral vein, basilic vein, and brachial vein. The videos will also include structures in close proximity to the intended veins. Using such database, we will run various vessel tracking and identification algorithms to evaluate their performance. Our ultimate goal is to develop an algorithm that will aid the ultrasound operator in identifying structures and differentiating between arteries and veins.

ELIGIBILITY:
Inclusion Criteria:

* The subjects will be any person age 18 and older who can legally consent to being scanned by ultrasound

Exclusion Criteria:

* No exclusion criteria shall be based on race, ethnicity, gender, pregnancy status, or HIV status

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-02; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Stetten, MD/PhD, Principal Investigator — University of Pittsburgh, Dept of Bioengineering
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Davies MJ, Cronin KD, Domaingue CM. Pulmonary artery catheterisation. An assessment of risks and benefits in 220 surgical patients. Anaesth Intensive Care. 1982 Feb;10(1):9-14. doi: 10.1177/0310057X8201000103. PMID 7065401
- [Background] Patel C, Laboy V, Venus B, Mathru M, Wier D. Acute complications of pulmonary artery catheter insertion in critically ill patients. Crit Care Med. 1986 Mar;14(3):195-7. doi: 10.1097/00003246-198603000-00005. PMID 3943335
- [Background] Knoblanche GE. Respiratory obstruction due to haematoma following internal jugular vein cannulation. Anaesth Intensive Care. 1979 Aug;7(3):286. No abstract available. PMID 495941
- [Background] Kua JS, Tan IK. Airway obstruction following internal jugular vein cannulation. Anaesthesia. 1997 Aug;52(8):776-80. doi: 10.1111/j.1365-2044.1997.177-az0310.x. PMID 9291764
- [Background] Shield CF 3rd, Richardson JD, Buckley CJ, Hagood CO Jr. Pseudoaneurysm of the brachiocephalic arteries: a complication of percutaneous internal jugular vein catheterization. Surgery. 1975 Aug;78(2):190-4. PMID 1098191
- [Background] Gobeil F, Couture P, Girard D, Plante R. Carotid artery-internal jugular fistula: another complication following pulmonary artery catheterization via the internal jugular venous route. Anesthesiology. 1994 Jan;80(1):230-2. No abstract available. PMID 8291718
- [Background] Applebaum RM, Adelman MA, Kanschuger MS, Jacobowitz G, Kronzon I. Transesophageal echocardiographic identification of a retrograde dissection of the ascending aorta caused by inadvertent cannulation of the common carotid artery. J Am Soc Echocardiogr. 1997 Sep;10(7):749-51. doi: 10.1016/s0894-7317(97)70119-6. PMID 9339427